CLINICAL TRIAL: NCT01202682
Title: Heart Rate Changes During Normal Activity, Exercise, and Sleep in Normal Healthy Subjects With and Without Epilepsy
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Shaun Comfort, MD, Study Project Manager
Other Study IDs: E-34
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2010-09

CONDITIONS: Healthy; Exercise
Keywords: Healthy subject exercise study
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to gather ECG data during normal activity, exercise, and sleep from normal subjects with or without well-controlled epilepsy. This normal subject data will serve as "true negative" (i.e., no seizure occurring) challenge data for testing cardiac based seizure detection algorithms.

DETAILED DESCRIPTION:
The purpose of this study is to gather ECG data during normal activity, exercise, and sleep from normal subjects with or without well-controlled epilepsy. This normal subject data will serve as "true negative" (i.e., no seizure occurring) challenge data for testing cardiac based seizure detection algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years or older and may be of either sex and of any race.
2. Subject must be in good general health, fully ambulatory, and able to complete the physical aspects of testing requirements.
3. Subject must be willing and able to complete informed consent and HIPAA authorization.
4. Subject may be diagnosed with epilepsy but must be well controlled on their regular treatment regimen.
5. Women of childbearing potential must have a negative urine pregnancy test.

Exclusion Criteria:

1. Subjects with skin abnormalities or conditions that would interfere with ECG electrode patch placement or cause subject discomfort with patch placement.
2. Subjects report history of allergies or sensitivity to adhesive tapes or patches.
3. Subjects with severe psychiatric disease that in the investigator's judgment would prevent the subject's successful completion of the study.
4. Subjects with epilepsy experiencing status epilepticus within the last 6 months.
5. Subjects with cardiovascular, respiratory, neuromuscular or gait disorders that in the investigator's judgment would cause unnecessary risk or inability to participate in the protocol.
6. Subjects with known cardiovascular arrhythmias or cardiac disease resulting in history of cardiac disease or abnormal ECG recordings. These include, but are not limited to, conditions such as chronic atrial fibrillation and permanent cardiac pacemaker implantation.
7. Use of beta adrenergic antagonists (i.e., "beta blockers") or calcium channel blocker agents that may affect heart rate.
8. Subjects currently dependent on alcohol or narcotic drugs as defined by DSM IV-TR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal, healthy population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials of Texas, San Antonio, Texas, United States